CLINICAL TRIAL: NCT06555159
Title: EFFECT OF AN AEROBIC EXERCISE PROGRAM ON METABOLIC DISORDERS LEVELS IN HIGHER EDUCATION STUDENTS AT THE UNIVERSITY OF COLIMA, RANDOMIZED CLINICAL TRIAL.
Brief Title: Exploring Physical Exercise for the Regulation and Control of Metabolic Disorders in College Students.
Acronym: (EPE_RCTMCS)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Colima (Other)
Collaborators: Pedro Julián Flores Moreno (Unknown); Nelson Enrique Ramos Cuevas (Unknown)
Responsible Party: Principal Investigator, Fabian Rojas Larios, Doctor en ciencias médicas, Universidad de Colima
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-6
Record Dates: First submitted 2024-08-12; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Metabolic Disorders; Abdominal Obesity; Blood Pressure Disorders; Hypertriglyceridemia; Hyperglycemia; HDL-Deficiency
Keywords: Exercise; Obesity; HDL; Triglycerides; Hypertension
MeSH Terms: conditions — Metabolic Diseases; Obesity, Abdominal; Hypertriglyceridemia; Hyperglycemia; Hypoalphalipoproteinemias; Motor Activity; Obesity; Hypertension | interventions — Jogging; Swimming

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants do not know if they belong to the control group or the experimental group Simple randomization will be performed using sealed envelopes, each containing a letter indicating group assignment that will not be seen by participants
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Continuous aerobic physical exercise program with progressive intensity loads (Experimental): Exercise prescription: jogging, swimming, and static cycling, three times a week with a duration of 60 minutes per exercise session with a progressive intensity, which will start at 57%-63% of the maximum heart rate (HRmax) in the first 4 weeks of the study, and will increase to 64% -76% in the final four weeks.
  Interventions: Behavioral: Physical exercise prescription: Continuous aerobic training (jogging, swimming, static cycling)
- Continuous aerobic physical exercise (Active Comparator): Intervention: Performing aerobic physical exercise: walking at 57% to 76% of HRmax.
  Interventions: Behavioral: Control group: Continuous aerobic physical exercise

INTERVENTIONS:
Behavioral: Physical exercise prescription: Continuous aerobic training (jogging, swimming, static cycling) — Aerobic physical exercise (APE) program involving jogging, swimming, and static cycling, with a progressive intensity, which will start at 57%-63% of the maximum heart rate. (HRmax) in the first 4 weeks of the study, and will increase to 64% -76% in the final four weeks, fulfilling the principle of progressive overload
  Arms: Continuous aerobic physical exercise program with progressive intensity loads
Behavioral: Control group: Continuous aerobic physical exercise — Control group -A-, will perform aerobic physical exercise, which will be walking at 57% to 76% of HRmax, keeping this intensity for the 8 week intervention period.
  Arms: Continuous aerobic physical exercise

SUMMARY:
This clinical trial objective is to evaluate the effect of an aerobic physical exercise program on reducing triglycerides, blood pressure, abdominal obesity, altered glucose levels, and the increase in HDL in college-level students at the University of Colima. It will try to answer whether aerobic physical exercise reduces metabolic disorders (altered blood pressure and glucose levels, abdominal obesity, and increased HDL). A simple randomized clinical trial will be conducted with a sample of 48 voluntary students from the University of Colima, divided into two groups of 24 people (Control group -A-, will perform aerobic physical exercise, which will be walking at 57% to 76% of HRmax; and Experimental Group -B-, will undergo an aerobic physical exercise (APE) program involving jogging, swimming, and static cycling, with a progressive intensity, which will start at 57%-63% of the maximum heart rate (HRmax) in the first 4 weeks of the study, and will increase to 64% -76% in the final four weeks, fulfilling the principle of progressive overload).

Researchers will compare the results of both groups to confirm the effectiveness of the planned aerobic physical exercise in reducing these risks.

DETAILED DESCRIPTION:
Once the project is approved by the Bioethics Committee from the Faculty of Medicine at the University of Colima and the Ethics Committee from Colima's Regional Hospital, annexing a no-conflict of interest letter, letters of intent will be prepared and sent to the directors of the faculties within the central campus of the University of Colima. Their purpose is to inform them about the project's generalities, obtain permission to share it with the students and address any questions they may have Those who agree will receive an informed consent form for their respective signatures. They will be informed about the appropriate attire for the study (for women, this includes sports shoes, leggings, and a top or T-shirt, and for men, shorts and a T-shirt), the requirement to fast for a minimum of 8 hours on the data collection day, and the date (Saturdays), time (8:00 am to 12:00 pm) and place (Faculty of Medicine, University of Colima) of the initial tests (these tests will also be considered the baseline for people who are found to have a metabolic alteration).

On assessment day, the project team will execute the following tests: application of the IPA-Q questionnaire, abdominal circumference, blood pressure, blood collection by venipuncture for HDL, triglycerides and glycemia, and the Queen's College step test to determine their cardiorespiratory capacity, (after completing all the tests, every participant will receive refreshments and will be asked if they are in good condition to conclude their assessments, if not, they will be monitored until their answer is affirmative).

Once all blood samples are collected, they will be taken to the laboratory at the Faculty of Chemical Sciences, University of Colima, for processing. Simultaneously, data from the other assessments will be synthesized. When the final results from all 5 tests are collected, a sample of 48 subjects will be selected for the protocol, considering the established inclusion criteria. With this sample, simple randomization will be performed in a new meeting, using sealed envelopes (each containing a letter indicating group assignment that will not be seen by participants). Participants will draw an envelope and mark it with their names, and they will hand the envelope to the designated person (principal investigator).

At the end of the meeting, the envelopes will be opened by the organizers in the absence of the participants to reveal whether they belong to the (A) control or (B) experimental group. This process ensures single-blind criteria, where participants do not know their group assignment.

After forming the (A) control and (B) experimental groups, they will be divided to provide them instructions for compliance with the exercise program while maintaining single-blind conditions. In the control group (A), the exercise prescription used by Habibzadeh in 2010 will be implemented: which involves walking for 30 minutes at an intensity of 57% to 76% of the maximum heart rate, three times per week (Monday, Wednesday, and Friday) for eight weeks. They will always be accompanied by a previously trained physical education student (Monitoring the intensity range in which the subjects must be during the session, will be done through the effort perception scale, heart rate at 15 seconds multiplied by 4 or the H10 polar monitor) (83). On the other hand, the experimental group (B) will engage in an aerobic exercise program (jogging, aquatic activities, and stationary cycling) lasting 40 to 60 minutes, three times per week (Monday, Wednesday, and Friday) for eight weeks, always under the supervision of the principal investigator. Each participant in the experimental group will receive a structured exercise prescription tailored to their specific condition, considering the established aerobic training ranges (57% to 63% of maximum heart rate). (Monitoring the intensity range in which the subjects must be during the session will be done through the effort perception scale, heart rate at 15 seconds multiplied by 4 or the H10 polar monitor).

By the end of the first four weeks, the second round of assessments and samples will be done, taking into consideration: Abdominal circumference, blood pressure), blood collection by venipuncture for HDL, triglycerides and glycemia, and the Queen's College step test will be performed (3 minutes), (after completing all the tests, every participant will receive refreshments and will be asked if they are in good condition to conclude their assessments, if not, they will be monitored until their answer is affirmative). Subsequently, after completing sample collection and assessments, the control group (A) will continue with the same dynamics as in the initial weeks. The experimental group (B) will maintain the same exercises (jogging, aquatic activities, and stationary cycling), but their intensity may be adjusted from 64% to 76% of the maximum heart rate if favourable results are obtained from the cardiorespiratory fitness test since this shows the level of evolution of the subject after the initial intervention and thus, the FITT-VP principle in exercise prescription would be fulfilled.

At the end of the last 4 weeks of the aerobic physical exercise program, the same sampling will be concluded; Abdominal circumference, arterial pressure, blood collection by venipuncture for HDL, triglycerides and glycemia, and the Queen's College step test will be performed (3 minutes) (after completing all the tests, every participant will receive refreshments and will be asked if they are in good condition to conclude their assessments, if not, they will be monitored until their answer is affirmative), finishing the proposed intervention protocol.

The statistical analysis will be conducted using the Statistical Package for the Social Sciences (SPSS) Statistics 26 from Business Machine (IBM). Descriptive statistics will be carried out, including measures of central tendency for the variables of age, sex and IPA-Q. Normality tests will be applied such as Kolmogorov-Smirnov for samples >50, and Shapiro-Wilk for samples <50. For the levels of triglycerides, glucose, HDL (High-Density Lipoprotein), abdominal circumference, and cardiorespiratory fitness, paired-sample T-tests will be used if the data follow a normal distribution, but if they do not, the Wilcoxon signed-rank test will be employed. To compare the control and experimental groups, independent-sample t-tests will be used if the data is normally distributed, otherwise the Mann-Whitney U test will be used. Likewise, a multivariate analysis will be carried out to relate the influence of physical exercise on metabolic alterations. A significance level of p ≤ 0.05 will be considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* University of Colima students linked to the central campus.
* Students aged between 18 and 25 years old.
* Authorization to participate in the project with a signed informed consent.
* Suffer from at least one of the parameters of metabolic disorders or cardiovascular risk (Hyperglycemia, decreased DHL, elevated triglycerides, abdominal obesity or hypertension) following the clinical assessment (Considering the criteria established by the ADA and ATPIII).

Exclusion Criteria:

* Motor limitations that may hinder the performance of physical exercise.
* Pregnancy or lactation.
* High Vigorous Physical Activity Level according to the IPA-Q.
* To be currently under pharmacological treatment to manage altered metabolic levels.

ELIMINATION CRITERIA

* Musculoskeletal injuries during the study period.
* Unforeseen Medical Events: Unexpected medical situations that could influence study results, such as hospitalizations, serious illnesses, or surgeries.
* Non-Compliance with Follow-Up: Subjects failing to meet a minimum of 80% (19 out of 24 sessions) of the stipulated physical conditioning program time.
* Initiation of clinical treatment that may affect protocol results, such as medications that reduce alterations.
* Participants who voluntarily withdraw from the study.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
HDL (Lipidic profile) | For the selected participants, this measurement will be taken a second time, after 4 weeks of exercise prescription, and a third time at the end of the protocol, after 8 weeks.
  Participants will undergo a blood extraction procedure during the test session, which will be in the care of a nurse to maximize the effectiveness of the procedure and reduce risks. Once all blood samples are collected, they will be taken to the laboratory at the Faculty of Chemical Sciences, University of Colima, for processing.
  If participants have any metabolic alterations (Males < 40 mg/dl, Females < 50 mg/dl), they will be considered candidates for this protocol.
hypertriglyceridemia | For the selected participants, this measurement will be taken a second time, after 4 weeks of exercise prescription, and a third time at the end of the protocol, after 8 weeks.
  Participants will undergo a blood extraction procedure during the test session, which will be in the care of a nurse to maximize the effectiveness of the procedure and reduce risks. Once all blood samples are collected, they will be taken to the laboratory at the Faculty of Chemical Sciences, University of Colima, for processing If participants have any metabolic alterations (Males >150 mg/dl; Females >150 mg/dl), they will be considered candidates for this protocol.
  For the selected participants, this measurement will be taken a second time, after 4 weeks of exercise prescription, and a third time at the end of the protocol, after 8 weeks.
Glucose alterations | For the selected participants, this measurement will be taken a second time, after 4 weeks of exercise prescription, and a third time at the end of the protocol, after 8 weeks.
  Participants will undergo a blood extraction procedure during the test session, which will be in the care of a nurse to maximize the effectiveness of the procedure and reduce risks. Once all blood samples are collected, they will be taken to the laboratory at the Faculty of Chemical Sciences, University of Colima, for processing If participants have any metabolic alterations (>110 mg/dl), they will be considered candidates for this protocol.
Arterial Hypertension | For the selected participants, this measurement will be taken a second time, after 4 weeks of exercise prescription, and a third time at the end of the protocol, after 8 weeks.
  Individuals have to remain seated for 5 to 10 minutes regulating their cardiorespiratory frequency. Afterwards, the clinician will start the measurement of blood pressure using a baumanometer. When the result is obtained, it will be corroborated using the cut-off points (Males > 130/85 mmHg Females > 130/85 mmHg), to determine the subject's participation
Abdominal circunference | At the beginning of the protocol, then 4 weeks later, and then 8 weeks later, when the intervention ends.
  For this test, a certified measuring tape will be used and it will also have the objective of determining the abdominal circumference taking into account the morphophysiological parameters established by the International Society for the Advancement of Kinanthropometry (ISAK) and a marker. The subject must be placed in an anatomical position and then will be told to raise his arms crossed at chest height. The upper edge of the iliac crest will be identified by marking it with the marker, and after that, the lower edge of the last rib will be identified, so a marking will be made, then the two established references will be taken to identify the middle area of the markings. The abdomen will be surrounded with the tape and the subject will be told to breathe normally, at the end of this, the circumference will be taken. If the subject has these measurements: Males >90cm and Females>85 cm, will be considered a study participant.
Queen College Step Test | At the beginning of the protocol, then 4 weeks later, and then 8 weeks later, when the intervention ends.
  This test aims to monitor the maximum oxygen consumption of the study subjects in 3 continuous minutes.
  At the end of the test, you will remain standing for 5 seconds, followed by taking the heart rate for 15 seconds, after which the partial result will be multiplied by 4 and the total result will be given.
  This result will be aligned with the percentiles of cardiorespiratory fitness, which range from 29.6 Vo2max to 42.4Vo2max in women and ranges from 34.1 Vo2max to 61 Vo2max in men, the lower the percentile, the lower the subject's cardiorespiratory capacity, which was aligned to determine your prescription for the exercise of the protocol.

SECONDARY OUTCOMES:
IPA Q questionnaire | Only at the beginning of the protocol
  The purpose of this questionnaire in its extended version, is to evaluate the level of physical activity of study participants during the last 7 days by minutes before completion.
  The total number of minutes will be added and the physical activity performed will be ranked either low, moderate or vigorous according to the guidelines determined by the WHO.

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Enrique Ramos Cuevas, BC, Principal Investigator — Universidad de Colima; Fabián Rojas Larios, PhD, Study Director — Universidad de Colima; Pedro Julián Flores, PhD, Study Director — Universidad de Colima
Locations (1):
- University of Colima, Colima, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kelley GA, Kelley KS, Tran ZV. Aerobic exercise and lipids and lipoproteins in women: a meta-analysis of randomized controlled trials. J Womens Health (Larchmt). 2004 Dec;13(10):1148-64. doi: 10.1089/jwh.2004.13.1148. PMID 15650348
- [Result] Silveira EA, Mendonca CR, Delpino FM, Elias Souza GV, Pereira de Souza Rosa L, de Oliveira C, Noll M. Sedentary behavior, physical inactivity, abdominal obesity and obesity in adults and older adults: A systematic review and meta-analysis. Clin Nutr ESPEN. 2022 Aug;50:63-73. doi: 10.1016/j.clnesp.2022.06.001. Epub 2022 Jun 14. PMID 35871953
- [Result] Sequi-Dominguez I, Alvarez-Bueno C, Martinez-Vizcaino V, Fernandez-Rodriguez R, Del Saz Lara A, Cavero-Redondo I. Effectiveness of Mobile Health Interventions Promoting Physical Activity and Lifestyle Interventions to Reduce Cardiovascular Risk Among Individuals With Metabolic Syndrome: Systematic Review and Meta-Analysis. J Med Internet Res. 2020 Aug 31;22(8):e17790. doi: 10.2196/17790. PMID 32865503
- [Result] Primo D, Garcia Rioja J, Izaola O, Del Rio San Cristobal C, Pinero Teno R, De Luis Roman D. [Real-world study of an online platform for the prescription of physical exercise to obese patients - Effect on anthropometric, biochemical parameters and quality of life]. Nutr Hosp. 2022 Mar 29;39(2):337-347. doi: 10.20960/nh.03842. Spanish. PMID 35068165
- [Result] Aristizabal JC, Montoya E, Sanchez YL, Yepes-Calderon M, Narvaez-Sanchez R, Gallo-Villegas JA, Calderon JC. Effects of Low-Volume, High-Intensity Interval Training Compared with Continuous Training on Regional and Global Body Composition in Adults with Metabolic Syndrome: A post hoc Analysis of a Randomized Clinical Trial. Ann Nutr Metab. 2021;77(5):279-288. doi: 10.1159/000518909. Epub 2021 Oct 6. PMID 34763335
- [Result] Alarcon-Gomez J, Chulvi-Medrano I, Martin-Rivera F, Calatayud J. Effect of High-Intensity Interval Training on Quality of Life, Sleep Quality, Exercise Motivation and Enjoyment in Sedentary People with Type 1 Diabetes Mellitus. Int J Environ Res Public Health. 2021 Nov 30;18(23):12612. doi: 10.3390/ijerph182312612. PMID 34886337
- [Result] Gallegos-Gonzalez G, Pineda-Garcia G, Serrano-Medina A, Martinez AL, Ochoa-Ruiz E. Association between Stress and Metabolic Syndrome and its Mediating Factors in University Students. Am J Health Behav. 2021 Nov 15;45(6):1091-1102. doi: 10.5993/AJHB.45.6.12. PMID 34969419

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT06555159/Prot_SAP_ICF_000.pdf
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-06-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT06555159/Prot_SAP_ICF_001.pdf